CLINICAL TRIAL: NCT06999733
Title: A Phase 1/2, Multicenter, Double-Masked, Placebo-Controlled Study of KB801 in Subjects With Stage 2 or 3 Neurotrophic Keratitis
Brief Title: A Study Assessing KB801 for the Treatment of Stage 2 or 3 Neurotrophic Keratitis
Acronym: EMERALD-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Krystal Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KB801-01
Record Dates: First submitted 2025-05-14; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Neurotrophic Keratitis
Keywords: Neurotrophic Keratitis; Persistent Corneal Epithelial Defect; Corneal Epithelial Defect

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- KB801 (Experimental)
  Interventions: Biological: KB801
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: KB801 — Ophthalmic suspension of replication-defective, non-integrating herpes simplex virus type 1 (HSV-1)-based vector delivering functional, full-length human nerve growth factor (NGF)
  Arms: KB801
Drug: Placebo — Vehicle
  Arms: Placebo

SUMMARY:
The Sponsor is developing KB801, a replication-defective, non-integrating herpes simplex virus type 1 (HSV-1)-derived vector engineered to deliver functional full-length human nerve growth factor (NGF) to the corneas of people with Stage 2 or 3 neurotrophic keratitis (NK) via topical application. This is a Phase 1/2, multicenter, double-masked, placebo-controlled study to evaluate the safety, tolerability, and preliminary efficacy of KB801 in these subjects.

DETAILED DESCRIPTION:
Subjects will will be randomized 2:1 to receive KB801 or placebo (vehicle) topically to the study eye twice weekly for 8 weeks. Subjects will return for follow-up visits 2- and 12-weeks after finishing treatment to monitor for safety and durability of corneal healing. Safety follow-up visits will then occur every 3 months up to 1 year on study.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have read, understood, and signed an Institutional Review Board (IRB) approved Informed Consent Form and must be willing and able to comply with study procedures and instructions.
2. Aged ≥ 18 years at the time of informed consent.
3. Diagnosis of Stage 2 or Stage 3 NK, as defined by the Mackie criteria.
4. Persistent corneal epithelial defect (PCED) of at least 2 weeks duration without clinical improvement during that time. PCED is defined as a focal loss of the cornea's outermost cell layer and can include involvement of the deeper stromal layers (i.e., corneal ulcer).
5. PCED at Screening 1 must have a minimum of 1 mm of any linear measurement of defect.
6. Decreased corneal sensitivity (≤ 4 cm using the Cochet-Bonnet esthesiometer [CBE]) within the area of the PCED and in at least one corneal quadrant outside of the area of the defect.
7. A negative pregnancy test at Screening 1 and Day 1 for women of child-bearing potential.

Exclusion Criteria:

1. An active ocular infection (bacterial, viral, fungal or protozoal) or active ocular inflammation not related to NK in the study eye as assessed by Investigator at Screening 1 or 2.
2. Use of any prohibited therapies at Screening or anticipated need for topical treatments other than the investigational product or products allowed per protocol in the study eye from Screening through the study Treatment Period

   1. The study Treatment Period is defined as Study Days 1 through 53
   2. Sufficient washout of prohibited therapies must occur prior to meeting eligibility criteria.
3. Anticipated use of therapeutic contact lenses or contact lens wear for refractive correction during the study Treatment Period in the study eye.
4. Evidence of corneal ulceration involving the posterior third of the corneal stroma, corneal melting, descemetocele, impending or perforation in the study eye at the time of Screening 1 or 2.
5. PCED at Screening 1 or 2 of > 8 mm maximum linear measurement in any eye.
6. The central 3 mm of corneas contain PCED bilaterally at Screening 1 or 2.
7. Anticipated need for punctal occlusion of the study eye during the Treatment Period.
8. Presence or history of any ocular or systemic disorder or condition that might hinder the efficacy of the study treatment or its evaluation, could possibly interfere with the interpretation of study results, or could be judged by the Investigator to be incompatible with the study visit schedule or conduct (e.g., progressive or degenerative corneal or retinal conditions, uveitis, optic neuritis, poorly controlled diabetes, autoimmune disease, systemic infection, neoplastic diseases).
9. Participation in another clinical study or treatment with an investigational agent 30 days or 5 half-lives, whichever is longer, prior to Day 1 (participation in a non-interventional observational study is permitted).
10. Intraocular surgery on the eligible eye(s) within 6 months prior to Screening 1, and any ophthalmic condition that may require surgery on the study eye during the Treatment Period. An exception to the preceding statement is allowed if, in the opinion of the Investigator, the ocular surgery is deemed the cause of the NK.
11. Corneal transplantation (i.e., keratoplasty) of the study eye. This includes full- or partial-thickness, or endothelial keratoplasty.
12. Subject who is pregnant or nursing.
13. Subject who is unwilling to comply with contraception requirements per-protocol (for subjects of childbearing potential).
14. Subject who is known to be noncompliant or is unlikely to comply with the requirements of the study protocol, in the opinion of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of KB801 based upon assessment of adverse events (frequency, severity, relatedness). | 8 weeks
  Number of subjects with treatment related adverse events as assessed by CTCAE v5.

SECONDARY OUTCOMES:
To evaluate the effect of KB801 on complete durable healing of the Persistent Corneal Epithelial Defect (PCED) in subjects with Stage 2 or Stage 3 NK | 10 weeks
  Proportion of subjects receiving KB801 with complete PCED closure at Week 8 AND Week 10 compared to those receiving placebo.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of California Irvine, Irvine, California
  - Azul Vision - California Eye Specialists Medical Group Inc., Pasadena, California
  - Midwest Cornea Associates, Carmel, Indiana
  - Vance Thompson Vision, Alexandria, Minnesota
  - Minnesota Eye Consultants, Minnetonka, Minnesota
  - UPMC Vision Institute, Pittsburgh, Pennsylvania